CLINICAL TRIAL: NCT06931366
Title: Outcomes of Internal Fixation of Tibial Plateau Fractures Involving Posterior Column According to Three Column Concept: Prospective Case Series
Brief Title: Posterior Column Fractures of Tibial Plateau
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Islam Abodeef Mahmoud Atia, Resident, Assiut University
Other Study IDs: 214117
Record Dates: First submitted 2025-04-09; First posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Tibial Plateau Fractures
MeSH Terms: conditions — Tibial Plateau Fractures | interventions — Open Fracture Reduction; Fracture Fixation, Internal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Open reduction and internal fixation — plates and screws

SUMMARY:
The goal of this observational study is to learn about the long-term effects of internal fixation methods in patients with posterior column fractures of tibial plateau according to three column concept. The main question it aims to answer is:

Does the internal fixation of posterior column fractures of tibial plateau according to three column concept has a good radiological and clinical outcomes in follow up for 1 year? Participants already having internal fixation for their posterior column fractures will do X ray in their follow up visit and answer survey questions about their joint pain, ROM for 1 year.

DETAILED DESCRIPTION:
The goal of this observational study is to measure the radiological and clinical long term effects of internal fixation methods in patients with posterior column fractures of tibial plateau according to three column concept by using Rasmussen score

ELIGIBILITY:
Inclusion Criteria:

* Skeletally mature patients (18 - 60 years old).
* Tibial plateau fracture with posterior column involvement classified by X-ray and CT scan
* Fractures within 3 weeks of trauma

Exclusion Criteria:

* Open fracture grade 3 Gustilo Anderson Classification but not managed by internal fixation within 3 weeks of trauma
* Paediatric fractures.
* Pathological fractures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Any public patient with posterior column tibial plateau fracture
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Anatomical reduction of articular surface of tibial plateau by Rasmussen score | From the enrollment to the end of treatment of 1 year
  This score measures the articular depression, condylar widening and angulation. Each result has a value which is summed all together where 18 is excellent, 12-17 is good, 6-10 is fair, less than 6 is poor

CONTACTS AND LOCATIONS:
Overall Officials: Ali F Abdelrahem, lecturer, Study Director — Department of Orthopedic Surgery and Traumatology, Assiut University; Aly M Mohamed, Prof, Study Chair — Department of Orthopedic Surgery and Traumatology, Assiut University
Locations (1):
- Assiut university trauma hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No